CLINICAL TRIAL: NCT00911248
Title: A Phase 2 Study to Assess the Efficacy, Safety, and Pharmacodynamic Activity of PTC299 in Patients With Neurofibromatosis Type 2
Brief Title: PTC299 for Treatment of Neurofibromatosis Type 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC299-ONC-007-NF2; NF080100
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Neurofibromatosis 2
Keywords: Angiogenesis; Neurofibromatosis; Post-transcriptional control; PTC299; VEGF
MeSH Terms: conditions — Neurofibromatosis 2; Neurofibromatoses | interventions — emvododstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTC299 (Experimental): PTC299 administered at 100 mg/dose twice per day
  Interventions: Drug: PTC299

INTERVENTIONS:
Drug: PTC299 — PTC299 will be administered orally at 100 mg/dose twice per day for up to 1 year or until tumor progression

SUMMARY:
Formation of new blood vessels (angiogenesis) is important for tumor growth in neurofibromatosis type 2 (NF2). It is known that tumors make a protein called vascular endothelial growth factor (VEGF) and there are higher levels of VEGF in the tumors and blood of many patients with NF2. VEGF stimulates the formation of blood vessels that supply the tumor with nutrients and oxygen. PTC299 is an oral drug that has been shown to decrease production of VEGF in animal models of human cancer. In these animal models, oral PTC299 administration decreases VEGF levels in the tumor and in the bloodstream, decreases blood vessel numbers in the tumor, and significantly slows or halts tumor growth. Safety studies in research animals indicate good tolerability at doses and drug levels that are higher than those planned for the clinical studies. Results from Phase 1a studies in healthy volunteers indicate that PTC299 achieves levels of PTC299 in the bloodstream that are known to be active in animal models of human tumor. This Phase 2 study is designed to test the hypothesis that PTC299 will be tolerable and will show evidence of VEGF reduction, antitumor activity, and hearing improvement when administered orally to patients with NF2.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages. In Stage 1 of the study, 11 patients will receive daily treatment with PTC299 administered at 100 mg/dose twice per day for up to 1 year or until tumor progression. If no subject responds with tumor shrinkage or an improvement in hearing, then the study will be stopped. If ≥1 out of 11 subjects respond, then the study will proceed to Stage 2 to enroll an additional 14 subjects for a total of 25 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of NF2
* Presence of vestibular schwannomas
* Evidence of progressive increase in vestibular schwannoma size or worsening hearing loss due to vestibular schwannoma
* Adequate functional status (Karnofsky Performance Score ≥60)
* Adequate bone marrow, liver, kidney function
* If sexually active, willingness to use effective barrier or medical contraception
* For women of childbearing potential, no pregnancy or breast-feeding
* Discontinuation of other therapies (except corticosteroids) for the treatment of NF2 and resolution of any acute toxic effects of prior therapies
* Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions
* Willingness to provide informed consent

Exclusion Criteria:

* Uncontrolled hypertension, major bleeding, HIV infection, or recent acute cardiovascular event
* Prior exposure to another anti-angiogenic therapy (eg, bevacizumab, sunitinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
To assess the effects of PTC299 on tumor volume and/or word recognition in patients with NF2. | 48 weeks

SECONDARY OUTCOMES:
To assess the effects of PTC299 on pure tone thresholds, brainstem auditory evoked responses (BAERs), and otoacoustic emissions (OAEs) in patients with NF2 | 48 weeks
To determine if PTC299 alters the perception of tinnitus | 48 weeks
To evaluate the effects of PTC299 on tumor blood flow | 48 weeks
To assess the effects of PTC299 on concentrations of circulating angiogenic factors or cytokines | 48 weeks
To describe the PTC299 safety profile | 48 weeks
To evaluate compliance with PTC299 treatment | 48 weeks
To assess PTC299 plasma exposure over time | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Barth, MD, Principal Investigator — PTC Therapeutics
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: PTC Therapeutics website — http://www.ptcbio.com